CLINICAL TRIAL: NCT01201096
Title: Neo-adjuvant Peptide Receptor Mediated Radiotherapy With 177Lutetium in Front of Curative Intended Liver Transplantation in Patients With Hepatic Metastasis of Neuroendocrine Tumors
Brief Title: Neo-adjuvant Peptide Receptor Mediated Radiotherapy With 177Lutetium in Front of Curative Intended Liver Transplantation in Patients With Hepatic Metastasis of Neuroendocrine Tumors (NEO-LEBE)
Acronym: NEO-LEBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Dr. med. Christine Wurst, Department of General-, Visceral- and Vascularsurgery, University of Jena
Other Study IDs: NEO-LEBE
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Liver; Metastasis; Neuroendocrine Tumors
Keywords: neuroendocrine tumor; liver metastasis; peptide receptor therapy; gastro-entero-pancreatic system
MeSH Terms: conditions — Neoplasm Metastasis; Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate; Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- peptide radioreceptor therapy and liver transplantation
  Interventions: Radiation: 177Lutetium; Procedure: Liver transplantation

INTERVENTIONS:
Radiation: 177Lutetium — two cycles of 177Lutetium radioreceptor therapy within two month
Procedure: Liver transplantation — about 9 month after finishing the receptor therapy liver transplantation takes place

SUMMARY:
The purpose of this study is to show the tumor free long term survival of patients with isolated non-resectable liver metastases of neuroendocrine tumors after neo-adjuvant radio receptor treatment and following liver transplantation.

DETAILED DESCRIPTION:
Matching patient will be treated neo-adjuvant at the hospital with 177 Lutetium peptide receptor radiotherapy in two following courses. After this treatment it will follow the liver transplantation within 9 month as postmortal or living donor liver transplantation.

Under certain conditions concerning the evaluation examinations patients can be included in the study.

Most important factors are no evidence of disease outside the liver, removed primary tumor, patients between 18 and 60 years, no curative surgical resection of the liver metastasis possible.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years
* neuroendocrine Tumor with low or intermediate malignant histological appearance
* primary tumor removed, no extrahepatic tumor
* liver metastasis not resectable
* positive evaluation for liver transplantation
* primary tumor drained by vena porta
* tumor load within the liver < 50%
* stable disease after receptor therapy with 177 Lutetium for 6 month

Exclusion Criteria:

* prognostic relevant second tumor disease
* pregnancy
* undifferentiated neuroendocrine carcinoma (WHO II, G3)
* renal insufficiency > second degree
* progressive carcinoid conditioned heart disease (>NYHA II)
* Karnofsky-Index < 60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients with liver metastasis of neuroendocrine tumors of the small bowel, colon, pancreas or stomach. Primary tumor removed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
tumor free survival | 5 years

SECONDARY OUTCOMES:
quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine Wurst, Dr. med., Principal Investigator — Department of general-, visceral- and vascular surgery, University of Jena; Dieter Hörsch, Prof. Dr. med, Study Director — Zentrum für neuroendokrine Tumore, Zentralklinik Bad Berka; Utz Settmacher, Prof. Dr. med., Study Chair — Department of general-, visceral- and vascular surgery, University of Jena; R. B. Baum, Prof.Dr.med., Principal Investigator — Center of neuroendocrine tumors, Zentralklinik Bad Berka
Locations (2):
- Germany (2):
  - Center for neuroendokrine tumors, Zentralklinik Bad Berka, Bad Berka, Thuringia
  - Department of general-, visceral- and vascular surgery, University of Jena, Jena, Thuringia